CLINICAL TRIAL: NCT02031653
Title: Comparison Between Invasive Pressure Flow Study and Non-invasive Penile Cuff Test
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, KYU-SUNG LEE, professor, Samsung Medical Center
Other Study IDs: 2013-07-151
Record Dates: First submitted 2014-01-08; First posted 2014-01-09 (Estimated); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Bladder Outlet Obstruction; Pressure Flow Study
Keywords: Penile Cuff Test
MeSH Terms: conditions — Urinary Bladder Neck Obstruction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study Group

SUMMARY:
To provide evidence of promising tests to noninvasively diagnose bladder outlet obstruction (BOO) in men with benign prostatic hyperplasia.

1. Penile cuff test provides a means of obtaining a urodynamic diagnosis with a high level of accuracy without the morbidity and expense of invasive Pressure flow study.
2. Penile cuff test may be particularly useful in the counseling of patients prior to benign prostatic hyperplasia operation. Patients diagnosed as obstructed following a penile cuff test can be reassured that surgery has a high chance of resulting in symptomatic benefit

ELIGIBILITY:
Inclusion Criteria:

1. Male patients with Low Urinary Tract Symptoms over 6 months. (International prostatic symptom score >= 12)
2. Patients scheduled to have pressure flow study.
3. Able to give fully informed consent

Exclusion Criteria:

1. Patients with urologic malignancies such as prostate cancer and bladder cancer
2. Patients underwent urethral, prostate surgery
3. Patients with urethral stricture or bladder diverticulum or bladder neck contracture
4. seems not to be appropriate to this study by the decision of investigators because of any other reasons

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients with Low Urinary Tract Symptoms over 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 335 (Actual)
Dates: Start 2014-01; Primary Completion 2017-07 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The Positive/Negative Predictive Value of Penile cuff test | 5 hours
The proportion comparison of Good responder between obstructed and unobstructed patients in penile cuff test | up to 3 months
  good responder: The reduction in the International Prostatic Symptom Scores of more than 50% from the initial scores 3 months after operation.

SECONDARY OUTCOMES:
The correlation of intra-vesical Pressure between Pressure flow study and penile cuff test | 5 hours
The difference of Pain visual analogue scale score between two diagnostic tests | 5 hours
The categorical change of penile cuff test normogram after BPH operation | up to 3 months
The PSA level change after benign prostatic hyperplasia operation in obstructed and non-obstructed patients. | up to 3 months .
The changes of International Prostatic Symptom Scores after BPH operation. | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea